CLINICAL TRIAL: NCT03299166
Title: A Randomized, Double-blind, Placebo-controlled Trial of Adjunctive Troriluzole in Obsessive Compulsive Disorder
Brief Title: Troriluzole (BHV-4157) in Adult Participants With Obsessive Compulsive Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV4157-202
Record Dates: First submitted 2017-09-28; First posted 2017-10-02 (Actual); Results first posted 2023-06-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Troriluzole (Experimental)
  Interventions: Drug: Troriluzole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Troriluzole — Troriluzole, 140 mg capsules once daily (QD) orally for the first 4 weeks and 200 mg (140 mg+ 60 mg capsules QD) for an additional 8 weeks
  Arms: Troriluzole
Drug: Placebo — Matching capsule once daily (QD)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of troriluzole as adjunctive therapy versus placebo in participants with obsessive compulsive disorder (OCD) who had an inadequate response to selective serotonin reuptake inhibitor (SSRI), clomipramine, venlafaxine, or desvenlafaxine treatment

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of OCD as per the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5).
2. Participants must be currently experiencing non-response or inadequate response to their current standard of care (SOC) medication defined as:

   1. Participant Yale-Brown Obsessive Compulsive Scale total score must be ≥ 19 at screening and Baseline, reflecting moderate or severe OCD symptoms.
   2. Participants must currently be on a SSRI, clomipramine, venlafaxine or desvenlafaxine.
3. Determined by the investigator to be medically stable at baseline/randomization as assessed by medical history, physical examination, laboratory test results, and electrocardiogram testing. Participants must be physically able and expected to complete the trial as designed;
4. Minimum of 6 years of education or equivalent and sufficiently fluent in English to complete necessary scales and understand consent forms;
5. Participants must have adequate hearing, vision, and language skills to perform neuropsychiatric testing and interviews as specified in the protocol;
6. Participants must be able to understand and agree to comply with the prescribed dosage regimens and procedures; report for regularly scheduled office visits; and reliably communicate with study personnel about adverse events and concomitant medications;
7. It is required that all women of child-bearing potential (WOCBP) who are sexually active agree to use two methods of contraception for the duration of the study (i.e. beginning 30 days prior to baseline and extending to 30 days after the last dose of study drug).
8. WOCBP must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to dosing at Baseline;
9. It is required that men who are sexually active with WOCBP agree to use 2 methods of contraception for the duration of the study (beginning at first treatment and extending to 90 days after the last dose of study drug).
10. The duration of the subject's OCD disease was to be ≥ 1 year.
11. In addition, subjects had to be on stable doses of other psychotropic medication for at least 12 weeks prior to screening.
12. Subjects had to have a Clinical Global Impression of Severity Scale (CGI-S) score of ≥ 4 at screening and baseline.

Exclusion Criteria:

1. Participants should be excluded with a history of more than 2 previous failed treatment trials of SSRIs, clomipramine, venlafaxine, or desvenlafaxine (not including the current SSRI trial) given for an adequate duration at an adequate dose as defined by the following criteria taken from the Massachusetts General Hospital Treatment Response Questionnaire for OCD (MGH-TRQ-OCD) as follows:

   1. Treatment failure / non-response: As per the MGH-TRQ-OCD, there has been minimal or no meaningful clinical benefit as perceived by the participant despite an adequate dose and duration of treatment;
   2. Adequate duration: At least 10 weeks of treatment with SSRI, clomipramine, venlafaxine, or desvenlafaxine
   3. Adequate dose: Defined by the the United States Prescribing Information labeling.
2. Evidence at screening or baseline of any medical or psychiatric condition other than OCD that could predominantly explain or contribute significantly to the subjects' symptoms or that could confound assessment of OCD symptoms
3. Mini Mental State Examination (MMSE) score of < 24 at Screening
4. Current or prior history, per DSM-5 criteria, of bipolar I or II disorder, schizophrenia or other psychotic disorders, schizoaffective disorder, autism or autistic spectrum disorders, borderline personality disorder, antisocial personality disorder, body dysmorphic disorder, hoarding disorder (symptoms of hoarding disorder as part of the OCD diagnosis are allowed, but a primary diagnosis of hoarding disorder is excluded); a current diagnosis of Tourette's disorder is also excluded;
5. Any eating disorder within the last 12 months;
6. Acute suicidality or suicide attempt or self-injurious behavior in the last 6 months;
7. History of psychosurgery, Deep Brain Stimulation (DBS) or Electroconvulsive Therapy (ECT).
8. Transcranial Magnetic Stimulation (TMS) is prohibited within 3 months prior to screening and during the study.
9. Participants who may have received a non-biological investigational agent in any clinical trial within 30 days, or a biological agent within 90 days prior to screening are excluded.
10. Creatinine ≥ 2 mg/dL.
11. Course of treatment for participants with localized cancers (without metastatic spread) is 5 years prior to screening.
12. QTcF (Fridericia) interval ≥ 470 msec during the screening or baseline period or uncontrolled arrhythmia or frequent premature ventricular contraction (PVCs) (> 5/minute) or Mobitz Type II second or third degree atrioventricular (AV) block or left bundle branch block, or right bundle branch block with a QRS duration ≥ 150 msec or intraventricular conduction defect with a QRS duration ≥150 msec or evidence of acute or sub-acute myocardial infarction or ischemia and added or other electrocardiogram findings that, in the investigator's opinion, would preclude participation in the study.
13. Previous treatment with riluzole

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2025-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (57):
- United States (57):
  - Metropolitan Neuro Behavioral Institute, Chandler, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - University of California San Diego, La Jolla, California
  - Synergy Research San Diego, Lemon Grove, California
  - CalNeuro Research Group, Los Angeles, California
  - Pacific Research Partners, LLC, Oakland, California
  - NRC Research Institute, Orange, California
  - Desert Valley Research, Rancho Mirage, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - Stanford University, Department of Psychiatry and Behavioral Sciences, Stanford, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Mountain View Clinical Research, Inc., Denver, Colorado
  - Institute of Living / Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - University of Florida Department of Psychiatry, Gainesville, Florida
  - Galiz Research, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - SIH Research, Inc, Kissimmee, Florida
  - Harmony Clinical Research, North Miami Beach, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - iResearch Savannah, Savannah, Georgia
  - Chicago Research Center, Chicago, Illinois
  - University of Chicago Department of Psychiatry & Behavioral Neuroscience, Chicago, Illinois
  - AMR-Baber Research, Inc, Naperville, Illinois
  - Phoenix Medical Research, Inc., Prairie Village, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Pharmasite Research, Inc., Pikesville, Maryland
  - McLean Hospital, Belmont, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - Michigan Clinical Research PC, Ann Arbor, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - ActivMed Practices and Research, Inc., Portsmouth, New Hampshire
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Integrative Clinical Trials LLC, Brooklyn, New York
  - Bio Behavioral Institute, Great Neck, New York
  - New York State Psychiatric Institute, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Baylor College of Medicine, Houston, Texas
  - Psychiatric Alliance of the Blue Ridge, Inc., Charlottesville, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 56 sites in the United States.
Pre-assignment Details: A total of 426 participants were enrolled, of which 248 participants were randomized in a 1:1: ratio to receive troriluzole (BHV-4157) or placebo. A total of 178 participants were not randomized due to withdrawal of consent, lost to follow-up, failed inclusion/exclusion criteria, or other reasons.
Groups:
- Troriluzole - Randomization Phase: Randomization phase (Weeks 1 through 12): Participants received troriluzole 140 mg capsules once daily (QD) orally for the first 4 weeks and 200 mg (140 mg+ 60 mg capsules QD) for an additional 8 weeks in the double-blind (DB) randomization phase.
- Placebo - Randomization Phase: Randomization phase (Weeks 1 through 12): Participants received troriluzole matching placebo capsules QD orally for up to 12 weeks in the DB randomization phase.
Period: Overall Study
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase
Started (Participants who were randomized.) | 124 | 124
Treated | 122 | 122
Modified Intent-to- Treat (mITT) Participants (Modified intent-to-treat (mITT) participants in the randomization phase included randomized participants who received at least 1 dose of blinded study drug and provided a non-missing baseline assessment and at least 1 non-missing post-baseline efficacy assessment.) | 115 | 117
Completed | 101 | 109
Not Completed | 23 | 15
Not completed — Adverse Event | 9 | 4
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Physician Decision | 1 | 1
Not completed — Sponsor Decision | 3 | 0
Not completed — Lost to Follow-up | 2 | 4
Not completed — Randomization Error | 0 | 1
Not completed — Subject unable to return due to COVID | 1 | 0
Not completed — Unable to complete Week 12 visit at site | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated participants in the randomization phase: Enrolled participants who received at least 1 dose of blinded study therapy (troriluzole or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase | Total
Number analyzed (Participants) | 122 | 122 | 244
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.9 (13.09) | 35.5 (13.26) | 36.7 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 74 | 149
  Male | 47 | 48 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 17 | 27
  Not Hispanic or Latino | 112 | 105 | 217
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 8 | 7 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 7 | 19
  White | 100 | 103 | 203
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Total Y-BOCS score at Randomization [Mean (Standard Deviation); unit: Units on a scale] — The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is a clinician-administered scale used extensively in research and clinical practice to both rate severity of obsessive compulsive disorder (OCD) and to monitor improvement during treatment. The scale consists of 10 items; the first 5 items assess obsessions, and the last 5 items assess compulsions. Subscale scores can be calculated for obsessions and compulsions, each on a scale of 0 to 20. A total score ranging from 0 to 40 can then be correlated to overall severity. The higher the number on the Y-BOCS, the more severe the symptoms.
  Units on a scale | 25.9 (3.91) | 26.0 (4.32) | 26.0 (4.11)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) Total Score
Description: The Y-BOCS is a clinician-administered scale used extensively in research and clinical practice to both rate severity of obsessive compulsive disorder (OCD) and to monitor improvement during treatment. It is designed to rate the severity of obsessions and compulsions as well as the type of symptoms in patients with OCD. The scale consists of 10 items; the first 5 items assess obsessions, and the last 5 items assess compulsions. Subscale scores can be calculated for obsessions and compulsions, each on a scale of 0 to 20. A total score ranging from 0 to 40 can then be correlated to overall severity. The higher the number on the Y-BOCS, the more severe the symptoms.
Time Frame: Baseline, Week 12
Population: mITT: Randomized participants who received at least 1 dose of study therapy and provided a non-missing baseline assessment and at least 1 non-missing post-baseline efficacy assessment in the randomization phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 115 | 117
Scores on a scale | -5.91 [-7.05 to -4.77] | -4.91 [-6.03 to -3.79]
Statistical Analysis 1: Comparison: Troriluzole - Randomization Phase vs Placebo - Randomization Phase; Model-based summary statistics are from a mixed model with repeated measures, including fixed effects for treatment, visit, treatment-by-visit interaction, baseline score, baseline score-by-visit interaction as covariates, and participant as random effect; Test type: Superiority; p = 0.2202, Mixed Models Analysis; LS Mean Difference = -1.00, 95% CI 2-sided [-2.59 to 0.60], Standard Error of Mean 0.81

2. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs) and AEs Leading to Study Drug Discontinuation in the DB Randomization Phase
Description: An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in participants or clinical investigation participants administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. An SAE was defined as any event that met any of the following criteria at any dose: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received study drug; other important medical events that may not have resulted in death, been life-threatening, or required hospitalization, or, based upon appropriate medical judgment, may have jeopardized the participant and may have required medical or surgical intervention to prevent other serious outcomes.
Time Frame: Up to 12 weeks
Population: Treated participants in the randomization phase
Measure: Number; unit: participants
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 122 | 122
participants
  Participants with at least 1 AE | 61 | 61
  Participants with at least 1 SAE | 0 | 0
  Participants with at least 1 AEs Leading to Study Drug Discontinuation | 13 | 5

3. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs) and AEs Leading to Study Drug Discontinuation in the Open-Label Extension Phase
Description: An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in participants or clinical investigation participants administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. An SAE was defined as any event that met any of the following criteria at any dose: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received study drug; other important medical events that may not have resulted in death, been life-threatening, or required hospitalization, or, based upon appropriate medical judgment may, have jeopardized the participant and may have required medical or surgical intervention to prevent other serious outcomes.
Time Frame: Up to 192 weeks
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities During the DB Randomization Phase
Description: Clinically significant laboratory abnormalities were defined as Grade 3 or 4 laboratory test results according to numeric laboratory test criteria found in Common Technical Criteria for Adverse Events Version 5.0 (2017) if available; otherwise, according to Division of Acquired Immune Deficiency Syndrome Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1 (2017). Laboratory tests of clinical interest for troriluzole included absolute neutrophil count < 500 per mm^3, alanine aminotransferase or aspartate aminotransferase > 3x upper limit of normal (ULN), and total bilirubin ≥ 2x ULN (Laboratory results were presented in US units).
Time Frame: Up to 12 weeks
Population: Treated participants in the randomization phase
Measure: Number; unit: participants
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 122 | 122
participants
  Hemoglobin, serum: number analyzed (Participants) | 119 | 118
  Hemoglobin, serum | 0 | 0
  Lymphocytes, low: number analyzed (Participants) | 119 | 117
  Lymphocytes, low | 0 | 0
  Lymphocytes, high: number analyzed (Participants) | 119 | 117
  Lymphocytes, high | 0 | 0
  Neutrophils: number analyzed (Participants) | 119 | 118
  Neutrophils | 0 | 1
  Platelets: number analyzed (Participants) | 119 | 118
  Platelets | 0 | 0
  White blood cells: number analyzed (Participants) | 119 | 118
  White blood cells | 0 | 0
  Alanine Aminotransferase: number analyzed (Participants) | 118 | 118
  Alanine Aminotransferase | 0 | 0
  Albumin: number analyzed (Participants) | 118 | 118
  Albumin | 0 | 0
  Alkaline Phosphatase: number analyzed (Participants) | 118 | 118
  Alkaline Phosphatase | 0 | 0
  Aspartate Aminotransferase: number analyzed (Participants) | 118 | 118
  Aspartate Aminotransferase | 2 | 0
  Bicarbonate: number analyzed (Participants) | 118 | 118
  Bicarbonate | 0 | 0
  Bilirubin: number analyzed (Participants) | 118 | 118
  Bilirubin | 0 | 0
  Calcium, low: number analyzed (Participants) | 118 | 118
  Calcium, low | 0 | 0
  Calcium, high: number analyzed (Participants) | 118 | 118
  Calcium, high | 0 | 0
  Creatine Kinase: number analyzed (Participants) | 118 | 118
  Creatine Kinase | 6 | 2
  Creatinine: number analyzed (Participants) | 118 | 118
  Creatinine | 0 | 0
  Glucose, Serum, low: number analyzed (Participants) | 118 | 118
  Glucose, Serum, low | 0 | 1
  Glucose, Serum, high: number analyzed (Participants) | 118 | 118
  Glucose, Serum, high | 0 | 0
  Lactate Dehydrogenase: number analyzed (Participants) | 118 | 118
  Lactate Dehydrogenase | 0 | 0
  Potassium, low: number analyzed (Participants) | 118 | 118
  Potassium, low | 0 | 0
  Potassium, high: number analyzed (Participants) | 118 | 118
  Potassium, high | 1 | 0
  Sodium, low: number analyzed (Participants) | 118 | 118
  Sodium, low | 0 | 1
  Sodium, high: number analyzed (Participants) | 118 | 118
  Sodium, high | 0 | 0
  Urate: number analyzed (Participants) | 118 | 117
  Urate | 0 | 0
  Glucose, Urine: number analyzed (Participants) | 119 | 118
  Glucose, Urine | 1 | 1
  Protein, Urine: number analyzed (Participants) | 119 | 118
  Protein, Urine | 0 | 0

5. Secondary Outcome: Change From Baseline in Functional Disability Assessed Using the Sheehan Disability Scale (SDS) Total Score
Description: The SDS was assessed in 3 domains: work/school (0-10), social life (0-10), and family life (0-10). The score from each domain was summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired). If the participant has not worked or studied for reasons unrelated to OCD, then the total score was considered as missing.
Time Frame: Baseline, Week 12
Population: The mITT participants in the randomization phase with available data were analyzed
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 102 | 105
Scores on a scale | -4.68 [-6.01 to -3.36] | -3.68 [-4.96 to -2.39]

6. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity Scale (CGI-S) Score
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline, Week 12
Population: mITT participants
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 115 | 117
Scores on a scale | -0.67 [-0.84 to -0.50] | -0.59 [-0.76 to -0.42]

7. Secondary Outcome: Change From Baseline in the Y-BOCS Obsessions Sub-Scale Score
Description: The Y-BOCS Obsessions Sub-scale consists of the last 5 items on the Y-BOCS and is measured on a scale of 0 to 20. A higher score on the Y-BOCS corresponds to greater symptom severity.
Time Frame: Baseline, Week 12
Population: mITT participants
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 115 | 117
Scores on a scale | -2.91 [-3.53 to -2.28] | -2.55 [-3.16 to -1.93]

8. Other Pre Specified Outcome: Change From Baseline in the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) Total Score at Weeks 4 and 8
Description: as for outcome 1
Time Frame: Baseline, Week 4 and Week 8
Population: mITT participants
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 115 | 117
Scores on a scale
  Week 4 | -3.40 [-4.26 to -2.53] | -2.93 [-3.78 to -2.08]
  Week 8 | -5.10 [-6.16 to -4.04] | -3.56 [-4.59 to -2.53]
Statistical Analysis 1: Comparison: Troriluzole - Randomization Phase vs Placebo - Randomization Phase; Week 4 Analysis. Model-based summary statistics are from a mixed model with repeated measures, including fixed effects for treatment, visit, treatment-by-visit interaction, baseline score, baseline score-by-visit interaction as covariates, and participant as random effect; Test type: Superiority; p = 0.4508, Mixed Models Analysis; LS Mean Difference = -0.46, 95% CI 2-sided [-1.67 to 0.75], Standard Error of Mean 0.61
Statistical Analysis 2: Comparison: Troriluzole - Randomization Phase vs Placebo - Randomization Phase; Week 8 Analysis. Model-based summary statistics are from a mixed model with repeated measures, including fixed effects for treatment, visit, treatment-by-visit interaction, baseline score, baseline score-by-visit interaction as covariates, and participant as random effect; Test type: Superiority; p = 0.0410, Mixed Models Analysis; LS Mean Difference = -1.54, 95% CI 2-sided [-3.02 to -0.06], Standard Error of Mean 0.75

ADVERSE EVENTS:
Time Frame: Randomization Phase: Maximum duration: 12 weeks
Description: Randomization phase: Treated participants in the randomization phase - enrolled participants who received at least 1 dose of blinded study therapy (troriluzole or placebo).
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/122
Other Adverse Events (participants affected / at risk) | 35/122 | 24/122
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Troriluzole - Randomization Phase (N=122) | Placebo - Randomization Phase (N=122)
Headache (Nervous system disorders) | 10 | 8
Dizziness (Nervous system disorders) | 9 | 2
Somnolence (Nervous system disorders) | 8 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 9
Nausea (Gastrointestinal disorders) | 8 | 2
Fatigue (General disorders) | 9 | 5
Nasopharyngitis (Infections and infestations) | 7 | 1

LIMITATIONS AND CAVEATS:
The provided results are from the DB Randomization Phase as the Open-Label Extension phase is still on-going.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT03299166/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT03299166/SAP_001.pdf